CLINICAL TRIAL: NCT04083326
Title: Digital Patient Journey Solution for Patients Undergoing Elective Hip and Knee Arthroplasty Due to Primary Osteoarthritis
Brief Title: Digital Patient Journey Solution for Patients Undergoing Elective Hip and Knee Arthroplasty Dueto Primary Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VTT Technical Research Centre of Finland (Other)
Collaborators: University of Oulu (Other); Oulu University Hospital (Other); Tampere University (Other); Buddy Healthcare Ltd (Unknown); Solteq Ltd (Unknown); Near Real Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Icory
Record Dates: First submitted 2019-08-29; First posted 2019-09-10 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Primary Elective Hip Arthroplasty (THA); Primary Elective Total Knee Arthroplasty (TKA)

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The group allocation is masked for the surgeon and for the outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Patient Journey Solution (Experimental): Patients in the intervention arm are provided with a digital patient journey solution used on a mobile device. The application is intended to be used during the whole care path. The patient can familiarize him-/herself to the phases of care through visual timeline representation of the care path, get information on how to prepare for a surgery, receive reminders, fill in questionnaire forms, communicate with the care personnel via messaging functionality and video calls, and search information from frequently asked questions. The application contains information about the preparation, forms for anamnesis, anesthesia and treatment follow-up, information videos and pictures, and timely and individually-tailored reminders, e.g., on when to stop eating and drinking before the surgery. In addition, the application provides instructions on how to arrive to the treatment unit and comprehensive guidance for wound care and rehabilitation at home after the operation.
  Interventions: Device: Digital Patient Journey Solution
- Conventional care group (No Intervention): Conventional care consists of specialist assessment in conjunction with pre-operative surgical visits and patient education. Patients in the conventional care group are provided with pre- and postoperative information face-to-face by paper-based method. Patients will be admitted and mobilised on the day of the surgery, and discharged one to three days after surgery. The follow-up visit, conducted by a physiotherapist, is conducted after 6 to 8 weeks post-discharge for patients with TKA and after 8 to 12 weeks for patients with THA.

INTERVENTIONS:
Device: Digital Patient Journey Solution — Patients in the intervention arm are provided with a digital patient journey solution used on a mobile device. The application is intended to be used during the whole care path. The patient can familiarize him-/herself to the phases of care through visual timeline representation of the care path, get information on how to prepare for a surgery, receive reminders, fill in questionnaire forms, communicate with the care personnel via messaging functionality and video calls, and search information from frequently asked questions. The application contains information about the preparation, forms for anamnesis, anesthesia and treatment follow-up, information videos and pictures, and timely and individually-tailored reminders, e.g., on when to stop eating and drinking before the surgery. In addition, the application provides instructions on how to arrive to the treatment unit and comprehensive guidance for wound care and rehabilitation at home after the operation.
  Arms: Digital Patient Journey Solution

SUMMARY:
This is an interventional study which aims at assessing the effects of a digital patient journey solution in patients undergoing elective hip and knee arthroplasty due to primary osteoarthritis.

DETAILED DESCRIPTION:
Traditionally, pre- and postoperative education has been provided face-to-face by paper-based methods for patients undergoing total hip arthroplasty (THA) and total knee arthroplasty (TKA). Digital patient journey solution has potential to enhance adherence to preoperative preparation and postoperative rehabilitation, and further improve patient experience, while reducing potential adverse events.

The purpose of this study is to assess a digital patient journey solution developed for patients undergoing elective hip and knee arthroplasty. The digital solution aims to support patient's preparation to and recovery from a hip and knee arthroplasty through provision of timely information and support related to preoperative preparation and postoperative rehabilitation. The information on the application is aligned with the patient's individual needs and requirements, and contains exercises to be completed daily for the duration of the program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing primary elective total hip or knee arthroplasty
* Diagnosis of primary osteoarthritis of hip or knee (M16.0, M16.1, M17.0, M17.1)
* Ability to speak, read and understand Finnish
* Access to a web-based device

Exclusion Criteria:

* Undergoing a total hip or knee arthroplasty revision
* A bilateral total hip or knee arthroplasty
* Total hip or knee arthroplasty following a rheumatoid arthritis
* Inability to walk with use of walking aids
* Unable to see or hear that impede the use of the digital patient journey solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Health-related quality of life measured with EuroQol EQ-5D-5L | Change from baseline up to 6-8 weeks after TKA or at 8-12 weeks after THA
  EuroQol EQ-5D-5L is a 5-level 5-dimensional standardized assessment tool. The index score (range 0-1 with 1 indicating perfect health and 0 indicating death) is used in the analyses.

SECONDARY OUTCOMES:
Change in the Western Ontario and McMaster Osteoarthritis Index (WOMAC) | Change from baseline up to 6-8 weeks after TKA or at 8-12 weeks after THA
  WOMAC is a disease-specific, self-administered health status instrument assessing pain, stiffness, and function in patients with osteoarthritis. Three subscale summary scores are used in the analysis: Pain (range:0-20), Stiffness (range: 0-8), Physical function (range 0-68) with lower scores indicating better health.
Patient experience post surgery | At discharge (1-3 days after the surgery)
  An 18-item questionnaire developed for the purposes of this study. The questionnaire entails 17 statements answered on a Likert scale and one open question for additional feedback. The questionnaire is compiled based on the following questionnaires: 11-scale by National Institute for Health and Welfare of Finland, NORPEQ, GS-PEQ and PPE- 15
Patient experience post intervention | 6-8 weeks after TKA or at 8-12 weeks after THA
  An 18-item questionnaire developed for the purposes of this study. The questionnaire entails 17 statements answered on a Likert scale and one open question for additional feedback. The questionnaire is compiled based on the following questionnaires: 11-scale by National Institute for Health and Welfare of Finland, NORPEQ, GS-PEQ and PPE- 15
Application user experience | 6-8 weeks after TKA or at 8-12 weeks after THA
  A 28-item questionnaire developed for the purposes of the study. The questionnaire includes questions with regard to, e.g., perceived usefulness, ease of use, ease of taking into use, and trust. The questions are drawn from Technology Acceptance Model for Mobile Services (TAMM). The questionnaire is asked from the intervention group only.
Technological self-efficacy | At baseline, and 6-8 weeks after TKA or at 8-12 weeks after THA
  Technological self-efficacy is measured with the Healthcare Technology Self-Efficacy (HTSE) -instrument adapted to the context of digital health services.
Self-efficacy regarding preoperative preparation | At baseline
  Self-efficacy is measured using a self-reported survey item developed for the purposes of this study.
Self-efficacy regarding postoperative preparation | At discharge (1-3 days after the surgery)
  Self-efficacy is measured using a self-reported survey item developed for the purposes of this study.
Self-efficacy during postoperative rehabilitation | At 1, 3, and 5 weeks after THA/TKA for the intervention group only
  Self-efficacy during rehabilitation is measured using self-reported survey items developed for the purposes of this study.
Change in Oxford Hip Score (OHS) | 60 days prior surgery and 120 days after the surgery
  OHS is a patient-reported outcome measure tool designed to assess disability in patients undergoing total hip replacement. The summary score (range: 12-60) is used in the analyses with higher scores indicating most difficulty. OHS is collected routinely as a part of the care path. For the study purposes these data are obtained post study from the existing medical records.
Change Oxford Knee Score (OKS) | 60 days prior surgery and 120 days after the surgery
  OKS is a patient-reported outcome measure tool designed to assess disability in patients undergoing total knee replacement. The summary score (range: 12-60) is used in the analyses with higher scores indicating most difficulty. OKS is collected routinely as a part of the care path. For the study purposes, these data are obtained post study from the existing medical records.
Preoperative adherence | From baseline until the date of the surgery for the intervention group only
  Percentage of completed instruction sheets (denominator is the number of all instruction sheets provided to the patient through the application)
Postoperative adherence | From discharge (1-3 days after the surgery) until 6-8 weeks after TKA or at 8-12 weeks after THA for the intervention group only
  The proportion of completed exercises (denominator is the number of all exercises provided to the patient through the application)

OTHER OUTCOMES:
Presurgical outpatient visits | From baseline until the date of the surgery. The data are collected post study from the existing medical records
  The number of presurgical outpatient visits
Cancellation of surgery | From baseline until the date of the surgery. The data are collected post study from the existing medical records
  Cancellation or postponement of surgery (yes/no)
Cancellation of postoperative follow-up visit | From the date of surgery until 6-8 weeks after TKA or at 8-12 weeks after THA. The data are collected post study from the existing medical records
  Cancellation or postponement of the postoperative follow-up visit (yes/no)
Hospital length of stay | From the date of surgery until hospital discharge (after the surgery). The data are collected post study from the existing medical records
  Hospital length of stay after TKA or THA (days)
Hospital readmission | From discharge (1-3 days after the surgery) until 6-8 weeks after TKA or at 8-12 weeks after THA. The data are collected post study from the existing medical records
  The number and date(s) for readmission(s) to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Minna Pikkarainen, PhD, Principal Investigator — University of Oulu
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No